CLINICAL TRIAL: NCT04161989
Title: The Effect of Omega 3 and Vaginal Progesterone on Birth Weight and Doppler Velocimetry of Constitutionally Small for Gestational Age Fetuses.
Brief Title: Omega 3 Plus Vaginal Progesterone on Birth Weight of Constitutionally Small for Gestational Age Fetuses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGA-VP
Record Dates: First submitted 2019-11-11; First posted 2019-11-13 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Small for Gestational Age at Delivery
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (omega-3 fatty acids group) (Other): received omega 3 (Omega 3 plus, SEDICO, Egypt); once daily from 28-30 weeks till delivery. The omega 3 plus capsule contains 1000 mg Fish Oil plus 100 mg Wheat Germ Oil is a natural source of Vitamin E.
  Interventions: Drug: omega-3 fatty acids
- Group II (vaginal progesterone plus omega-3 group) (Other): received vaginal progesterone (Prontogest 400 mg vaginal suppository, Marcyrl Pharmaceutical Industries, Egypt) and omega 3 once daily from 28-30 weeks till delivery.
  Interventions: Drug: omega-3 fatty acids; Drug: vaginal progesterone

INTERVENTIONS:
Drug: omega-3 fatty acids — . The Omega 3 plus capsule contains 1000 mg Fish Oil (contains Eicosapentaenoic acid 13% & Docosahexaenoic acid 9%) plus 100 mg Wheat Germ Oil (Linoleic acid 52- 59%) as a natural source of Vitamin E.
Drug: vaginal progesterone — Prontogest 400 mg vaginal suppository contains progesterone 400 mg.
  Arms: Group II (vaginal progesterone plus omega-3 group)

SUMMARY:
Small for gestational age refers to an infant born with a birth weight less than the 10th centile. Severe small for gestational age refers to an infant born with a birth weight less than the 3rd centile. Constitutionally small fetuses are fetuses whose growth at all gestational ages has been low but otherwise healthy. Those babies have a great risk for perinatal morbidity and mortality. Many causes are responsible for the development of Severe small for gestational age, however; in a few cases, the cause could not be detected. In contrast to pathologic intrauterine growth restriction, the constitutionally small fetuses have normal umbilical and middle cerebral artery Doppler velocimetry and normal amniotic fluid volume. In this circumstance, continued biophysical testing and delivery at 38-39 weeks is reasonable. Low birth weight fetuses comprise both preterm births and SGA. They are at a higher risk of adverse birth outcomes. So the trials to increase the blood flow to the uterus and/or the fetus may improve the neonatal outcomes. There are many lines of treatment that have been emerged now for the treatment of small for gestational age fetuses like maternal rest and oxygenation, aspirin therapy, supplementation of zinc, and fish oil. However; all mentioned lines of treatment lack evidence of effectiveness in literature. Omega-3 fatty acids as antioxidants inhibit the free radicals released during pregnancy which are responsible for vasoconstriction; so vasodilatation will occur. This leads to increase blood flow to the uterus and placenta which improves pregnancy outcomes. Progesterone is a smooth muscle relaxant and has a vasodilator effect on the blood vessels. It causes endothelium- relaxation of human placental arteries and veins. This relaxation is significant for maintaining low flow impedance and satisfactory blood flow in the placental circulation. DeFranco et al observed that vaginal progesterone is associated with vascular relaxation and increased uterine blood flow. But, he did not observe this vascular effect in women receiving systemic progesterone. So from the above evidence; there is a need to study the effect of omega 3 and progesterone on pregnant women whose pregnancy is complicated with constitutionally small for gestational age fetuses in trial to find a new line of treatment of this problem.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women aged 20-35 years.
2. Pregnant women from 28 to 30 weeks gestation.
3. Women with small for gestational age fetus. It refers to an estimated fetal weight or abdominal circumference <10th centile with no pathology is present.
4. Women with normal resistant index in uterine arteries at the time of recruitment.
5. Women with normal resistant index in umbilical arteries at the time of recruitment.

Exclusion Criteria:

1. Women with estimated fetal weight below the 5th or 3rd percentile.
2. Women with any major risk factors for intrauterine growth restriction.
3. Women with multiple pregnancies.
4. Women with low amniotic fluid volume or premature pre-labor rupture of membranes.
5. Women with antepartum hemorrhage or fetal congenital anomalies.
6. Women with absent or reversed diastolic flow in the umbilical artery at the time of recruitment.
7. Women with any contraindications for progesterone or omega 3.
8. Women who refused to participate in our study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
The difference in mean birth weight (gram) | 6 weeks

SECONDARY OUTCOMES:
Estimated fetal weight (gram) | 6 weeks
Time of delivery (weeks) | 6 weeks
Doppler indices in the umbilical artery | 6 weeks
Doppler indices in the uterine artery | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided